CLINICAL TRIAL: NCT01050075
Title: A Pilot Study Investigating the Feasibility of Using Acupuncture for the Treatment of Taxane-Induced Peripheral Neuropathy
Brief Title: Acupuncture in Treating Nerve Pain in Patients With Stage I, Stage II, or Stage III Breast Cancer Who Are Receiving Paclitaxel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit patients in the 6 month extension allowed.
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09109; NCI-2010-00103
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: male breast cancer; neurotoxicity; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Neurotoxicity Syndromes | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive paclitaxel as standard of care every 2 weeks for 4 courses. Patients undergo acupuncture therapy comprising 2 30-minute sessions a week for 4 weeks during courses 3 and 4.
  Interventions: Other: acupuncture therapy; Other: questionnaire administration; Other: management of therapy complications
- Arm II (Experimental): Patients receive paclitaxel as standard of care every 2 weeks for 4 courses. Patients then undergo acupuncture therapy comprising 2 30-minute sessions a week for 4 weeks.
  Interventions: Other: acupuncture therapy; Other: questionnaire administration; Other: management of therapy complications

INTERVENTIONS:
Other: acupuncture therapy — acupuncture therapy
  Other Names: acupuncture
Other: questionnaire administration — Ancillary study
Other: management of therapy complications — To be determined by the treating physician
  Other Names: complications of therapy, management of

SUMMARY:
RATIONALE: Acupuncture may help relieve nerve pain caused by chemotherapy.

PURPOSE: This randomized clinical trial is studying how well acupuncture works in treating nerve pain in patients with stage I, stage II, and stage III breast cancer who are receiving paclitaxel.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To explore the potential for the use of acupuncture to prevent a worsening of the nerve damage in patients (during treatment) due to paclitaxel as measured by a Neuropathic Pain Symptom Inventory.

SECONDARY OBJECTIVES:

I. Evaluate the impact of acupuncture based on neurological assessment, quantitative sensory tests and nerve conduction tests.

II. Evaluate the improvement observed when treating patients for peripheral neuropathy (post-chemotherapy) with acupuncture based on the same metrics.

III. To correlate objective measures of neuropathy (nerve conduction, quantitative sensory tests, neuropathy composite score, and blood cytokine levels) with the subjective questionnaire/quality of life measures.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel every 2 weeks for 4 courses as standard of care. Patients undergo acupuncture therapy comprising 2 30-minute sessions a week for 4 weeks during courses 3 and 4.

ARM II: Patients receive paclitaxel every 2 weeks for 4 courses as standard of care. Patients then undergo acupuncture therapy comprising 2 30-minute sessions a week for 4 weeks.

ELIGIBILITY:
Inclusion

* Patients must have a history of histologically or cytologically confirmed stage I, II, or III breast cancer that have received 2 cycles of paclitaxel, and expected to receive paclitaxel for two more cycles, and are experiencing grade 1 peripheral neuropathy (CTCAE criteria)
* Performance ECOG 0-2 (Karnofsky Performance Status >= 60%)
* Life expectancy of greater than 6 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion

* Patients with radiologically confirmed stage IV breast cancer
* Patients who had acupuncture in the previous 8 weeks
* Change in use of any of the following drugs in the prior 4 weeks: opiates, antidepressants, or anxiolytics ("change" is defined as initiation or cessation of treatment, or change in prescribed dose or regimen)
* Patients with needle phobia
* Patients who experienced any peripheral neuropathy prior to chemotherapy
* Patients who have the potential for serious bleeding due to inherited diseases such as hemophilia
* Patients with diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in the Neuropathic Pain Symptom Inventory Scores | At the end of 4 courses of chemotherapy

SECONDARY OUTCOMES:
Percentage of patients requiring a dose reduction or additional neuropathy distress related pharmacologic management | Eight weeks after study enrollment
Impact of assigning patients the worst score when dose reducing/or prescribing additional treatment | Eight weeks after study enrollment
Observed improvement in patients following treatment with acupuncture as to compared to those no longer receiving acupuncture | Eight weeks after study enrollment
Comparison of changes in neurological assessment of patients | At the end of therapy and 1 month after the end of therapy
Correlation between nerve inventory questionnaires and quantitative nerve tests | Eight weeks after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Harry Openshaw, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - City of Hope Medical Group Inc, Pasadena, California